CLINICAL TRIAL: NCT00071604
Title: Medication Adherence in Older Psychotic People
Brief Title: Medication Adherence in Older People With Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: R01MH062849 (NIH); R01MH062849 (NIH); DATR A4-GPS
Record Dates: First submitted 2003-10-29; First posted 2003-10-30 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2008-04

CONDITIONS: Psychotic Disorders; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

INTERVENTIONS:
Behavioral: Medication Adherence Therapy
Behavioral: Friendly Support Group

SUMMARY:
This study will determine whether Medication Adherence Therapy (MAT) can improve medication adherence and lower the risk of rehospitalization in older patients with psychosis.

DETAILED DESCRIPTION:
Psychoses are among the most common and serious psychiatric disorders. Currently, the most effective treatment for psychoses involves the use of antipsychotic or neuroleptic medications. Unfortunately, pharmacologic regimens often do not achieve their goals because of poor medication adherence. Nonadherence to antipsychotic treatment is a considerable public health problem that leads to myriad clinical and economic burdens, including psychotic relapse, increased clinic and emergency room visits, and rehospitalization.

Participants in this study are randomly assigned to receive either MAT or supportive treatment for 12 weeks. MAT is given in 15 sessions and consists of motivational interviewing, education, and social skills and behavior modification. Individual MAT sessions are held in Weeks 1 and 12; small group sessions take place in Weeks 2 through 11. Three monthly booster group sessions begin in Week 16. Participants are assessed at baseline and at 3, 6, and 12 months. Medication adherence, psychopathology, quality of life, medication side effects, health beliefs, and functioning are assessed.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for schizophrenia or schizoaffective disorder
* Outpatient status at the time of enrollment
* Currently prescribed maintenance treatment with antipsychotic medication (typical or atypical, oral or depot)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2002-09; Study Completion 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lacro, PharmD, Principal Investigator — VA San Diego Healthcare System & University of California, San Diego
Locations (1):
- Division of Geriatric Psychiatry Center (University of California, San Diego), San Diego, California, United States